CLINICAL TRIAL: NCT03638271
Title: Role of Cardiac Magnetic Resonance in Non Ischemic Cardiomyopathy
Brief Title: Cardiac Magnetic Resonance in Non Ischemic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Reham Sameeh (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Reham Sameeh, Assisstant lecturer, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Non ischemic cardiomyopathy MR
Record Dates: First submitted 2018-06-20; First posted 2018-08-20 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2020-10

CONDITIONS: Cardiac Magnetic Resonance Imaging in Non Ischemic Cardiomyopathy

STUDY DESIGN:
Intervention Model Description: prospective manner study will include 50 patients of both sex and different age with any type of cardiomyopathy diagnosed clinically or by Doppler echocardiography, will undergo cardiac magnetic resonance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nonischemic cardiomyopathic patient (Other): Patients in different sex and age groups diagnosed with any type of nonischemic cardiomyopathy clinically or with echocardiography will undergo cardiac magnetic resonance imaging.
  Interventions: Diagnostic Test: Cardiac magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Cardiac magnetic resonance imaging — Patients in different sex and age groups diagnosed with any type of nonischemic cardiomyopathy clinically or with echocardiography will undergo cardiac magnetic resonance imaging and compare their results.

SUMMARY:
Cardiac magnetic resonance imaging has been established as a promising three dimensional imaging modality with the ability to assess cardiac morphology, ventricular function, perfusion, viability and imaging characteristics of the surrounding vasculature without ionizing radiation. The accurate treatment of patients with cardiac disorders has created the need for accurate and reproducible measurements of cardiac chamber volumes and function. Cardiac magnetic resonance has the ability to provide this information as well as assess edema, perfusion, viability and vascular anatomy.

DETAILED DESCRIPTION:
Nonischemic cardiomyopathy is considered as a variety of structural and functional myocardial disorders in which the myocardium is abnormal in the absence of diseases such as hypertension and coronary artery, valvular, and congenital heart diseases. Classification of cardiomyopathies is complex, with many available systems. The American Heart Association broadly divides them into primary and secondary types. The European Society of Cardiology classifies cardiomyopathies into several distinct morphologic and functional phenotypes, each of which can be further subclassified into familial and nonfamilial forms . There is an overlap between genetic and acquired cardiomyopathies, especially in the category of dilated cardiomyopathies.

Cardiomyopathy has a prevalence of 0.02% of the population with annual death rates up to 25,000 in the United States. Nonischemic cardiomyopathy is more common in younger individuals and women.

Although echocardiography is the simplest imaging technique used for screening, diagnosis and classification of cardiomyopathies on the basis of morphology, it is operator dependent , has no tissue characterization capabilities and limited field of view especially in obese/chronic obstructive pulmonary disease patients, influenced by acoustic window, is not adequate in the evaluation of the right ventricle or extra-cardiac associated chest manifestations where magnetic resonance is superior in this issue . Transesophageal echocardiography has a better acoustic window, but it is an invasive procedure.

In comparison, cardiac multidetector computed tomography is less useful for the assessment of such cases currently because multidetector computed tomography involves radiation exposure and contrast medium- related problems and provides less information (ie, hemodynamic information, tissue characterization such as fibrosis) than magnetic resonance imaging does. Computed tomography would be more appropriate in specific requests to detect coronary calcification, exclude coronary artery disease and in those cases with contraindications for magnetic resonance imaging, such as a pacemaker.

Cardiac magnetic resonance imaging has been established as the best three dimensional imaging modality with the ability to assess cardiac morphology, ventricular function, perfusion, viability and imaging characteristics of the surrounding vasculature without ionizing radiation. The accurate treatment of patients with cardiac disorders has created the need for accurate and reproducible measurements of cardiac chamber volumes and function. Cardiac magnetic resonance has the ability to provide this information as well as assess oedema, perfusion, viability and vascular anatomy.

The high soft-tissue contrast, availability of a large field of view, multiplanar acquisition capability and lack of ionizing radiation are particularly appealing features of Cardiac magnetic resonance.

There are certain technical challenges unique to cardiac magnetic resonance image as rapid and complex motion of the heart and pulsations of the surrounding great vessels. In addition, the effects of respiratory motion and systolic ventricular blood velocities up to 200 cm/s further complicate cardiac imaging. These challenges are generally solved by implementation of electrocardiography (cardiac) gating; navigator echo respiratory gating; breath-hold techniques; rapid, high-performance gradients; improved field homogeneity; and advanced pulse sequences. electrocardiography gating can be either prospective or retrospective.

Several Cardiac magnetic resonance sequences are available for the evaluation of Nonischemic cardiomyopathy, each providing specific information. Depending on the clinical suspicion, the cardiac imager can add specific sequences to form a Cardiac magnetic resonance protocol tailored to that particular disease process.

Delayed myocardial enhancement, being one of cardiac magnetic resonance imaging sequences, is not specific for myocardial infarction and can be used in many other cardiac diseases. Delayed enhancement in nonischemic myocardial disease generally, unlike in ischemic heart disease, has no particular coronary artery distribution and is often midwall rather than subendocardial or transmural . Moreover, in the acute phase, the first-pass perfusion study usually does not show any focal perfusion defect in nonischemic cardiomyopathy but instead may show normal results or early increased enhancement.

Cardiac magnetic resonance has now established itself as a crucial imaging technique in the evaluation of several cardiomyopathies. It not only provides comprehensive information on structure and function, but also can perform tissue characterization, which helps in establishing the etiology of cardiomyopathy. Cardiac magnetic resonance is also useful in establishing the diagnosis, providing guidance for endomyocardial biopsy, accurate quantification of function, volumes, and fibrosis, prognostic determination, risk stratification, and monitoring response to therapy.

One of the most important added points in in investigator(s) research is to assess extra cardiac chest manifestation in by one session of magnetic resonance imaging session with high accuracy and least cost.

Echocardiography is the best available gold standard for cardiomyopathic patient as in multiple previous studies, so it well be done for each patient in investigator(s) study for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients in different sex and age groups with any type of cardiomyopathy and others non cardiomyopathic cases

Exclusion Criteria:

* Non compatible implantable devices with magnetic resonance machine in some cases as presence of anti para-magnetic substance as pacemakers.
* In severely ill patients as severe renal impairment (risk of nephrogenic systemic fibrosis)
* Those with sever claustrophobia.
* Dysrhythmia affecting ECG-gating.
* Early pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac morphological measurements. | Within two year
  Detection of cardiac wall thickness and ventricular systolic/diastolic diameters. all these measures in millimeters using cardiac magnetic resonance and compare results with echocardiography.
Cardiac contractility of each part | Within two year
  Visual assessment of cardiac motility in term of normo- , hypo-, or dys-kinesia using cardiac magnetic resonance and compare results with echocardiography.
Measurements of severity and prognosis of nonischemic cardiomyopathic patients | Within two year
  Detection of cardiac muscle replacement and fibrosis by delayed myocardial enhancement using cardiac magnetic resonance, which is indicator of severity and prognosis of disease.
Assessment of cardiac function. | Within two years
  Calculation of ejection fraction in percentage.

SECONDARY OUTCOMES:
Diagnosis and differentiation of different types of non-ischemic cardiomyopathic types. | Within two years
  Diagnosis and differentiation of different types of non-ischemic cardiomyopathic types according to previous measures.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Sameeh, assistant lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Elliott P, Andersson B, Arbustini E, Bilinska Z, Cecchi F, Charron P, Dubourg O, Kuhl U, Maisch B, McKenna WJ, Monserrat L, Pankuweit S, Rapezzi C, Seferovic P, Tavazzi L, Keren A. Classification of the cardiomyopathies: a position statement from the European Society Of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2008 Jan;29(2):270-6. doi: 10.1093/eurheartj/ehm342. Epub 2007 Oct 4. PMID 17916581
- [Background] Maron BJ, Towbin JA, Thiene G, Antzelevitch C, Corrado D, Arnett D, Moss AJ, Seidman CE, Young JB; American Heart Association; Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; Council on Epidemiology and Prevention. Contemporary definitions and classification of the cardiomyopathies: an American Heart Association Scientific Statement from the Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; and Council on Epidemiology and Prevention. Circulation. 2006 Apr 11;113(14):1807-16. doi: 10.1161/CIRCULATIONAHA.106.174287. Epub 2006 Mar 27. PMID 16567565
- [Background] Fuster V, Kim RJ. Frontiers in cardiovascular magnetic resonance. Circulation. 2005 Jul 5;112(1):135-44. doi: 10.1161/01.CIR.0000155618.37779.A0. No abstract available. PMID 15998698
- [Background] O'Donnell DH, Abbara S, Chaithiraphan V, Yared K, Killeen RP, Martos R, Keane D, Cury RC, Dodd JD. Cardiac MR imaging of nonischemic cardiomyopathies: imaging protocols and spectra of appearances. Radiology. 2012 Feb;262(2):403-22. doi: 10.1148/radiol.11100284. PMID 22282181
- [Background] Follath F. Nonischemic heart failure: epidemiology, pathophysiology, and progression of disease. J Cardiovasc Pharmacol. 1999 Jun;33 Suppl 3:S31-5. doi: 10.1097/00005344-199906003-00004. PMID 10442682
- [Background] WRITING COMMITTEE MEMBERS; Yancy CW, Jessup M, Bozkurt B, Butler J, Casey DE Jr, Drazner MH, Fonarow GC, Geraci SA, Horwich T, Januzzi JL, Johnson MR, Kasper EK, Levy WC, Masoudi FA, McBride PE, McMurray JJ, Mitchell JE, Peterson PN, Riegel B, Sam F, Stevenson LW, Tang WH, Tsai EJ, Wilkoff BL; American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. 2013 ACCF/AHA guideline for the management of heart failure: a report of the American College of Cardiology Foundation/American Heart Association Task Force on practice guidelines. Circulation. 2013 Oct 15;128(16):e240-327. doi: 10.1161/CIR.0b013e31829e8776. Epub 2013 Jun 5. No abstract available. PMID 23741058
- [Background] Williams TJ, Manghat NE, McKay-Ferguson A, Ring NJ, Morgan-Hughes GJ, Roobottom CA. Cardiomyopathy: appearances on ECG-gated 64-detector row computed tomography. Clin Radiol. 2008 Apr;63(4):464-74. doi: 10.1016/j.crad.2007.07.024. Epub 2007 Nov 5. PMID 18325368
- [Background] Pohost GM. The history of cardiovascular magnetic resonance. JACC Cardiovasc Imaging. 2008 Sep;1(5):672-8. doi: 10.1016/j.jcmg.2008.07.009. No abstract available. PMID 19356498
- [Background] Marwick TH, Schwaiger M. The future of cardiovascular imaging in the diagnosis and management of heart failure, part 1: tasks and tools. Circ Cardiovasc Imaging. 2008 Jul;1(1):58-69. doi: 10.1161/CIRCIMAGING.108.792408. No abstract available. PMID 19808515
- [Background] Boxt LM. Cardiac MR imaging: a guide for the beginner. Radiographics. 1999 Jul-Aug;19(4):1009-25; discussion 1026-8. doi: 10.1148/radiographics.19.4.g99jl161009. PMID 10464806
- [Background] Reeder SB, Du YP, Lima JA, Bluemke DA. Advanced cardiac MR imaging of ischemic heart disease. Radiographics. 2001 Jul-Aug;21(4):1047-74. doi: 10.1148/radiographics.21.4.g01jl281047. PMID 11452080
- [Background] Scott AD, Keegan J, Firmin DN. Motion in cardiovascular MR imaging. Radiology. 2009 Feb;250(2):331-51. doi: 10.1148/radiol.2502071998. PMID 19188310
- [Background] American College of Cardiology Foundation Task Force on Expert Consensus Documents; Hundley WG, Bluemke DA, Finn JP, Flamm SD, Fogel MA, Friedrich MG, Ho VB, Jerosch-Herold M, Kramer CM, Manning WJ, Patel M, Pohost GM, Stillman AE, White RD, Woodard PK. ACCF/ACR/AHA/NASCI/SCMR 2010 expert consensus document on cardiovascular magnetic resonance: a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents. J Am Coll Cardiol. 2010 Jun 8;55(23):2614-62. doi: 10.1016/j.jacc.2009.11.011. No abstract available. PMID 20513610
- [Background] McCrohon JA, Moon JC, Prasad SK, McKenna WJ, Lorenz CH, Coats AJ, Pennell DJ. Differentiation of heart failure related to dilated cardiomyopathy and coronary artery disease using gadolinium-enhanced cardiovascular magnetic resonance. Circulation. 2003 Jul 8;108(1):54-9. doi: 10.1161/01.CIR.0000078641.19365.4C. Epub 2003 Jun 23. PMID 12821550
- [Background] Rajiah P, Raza S, Saboo SS, Ghoshhajra B, Abbara S. Update on the Role of Cardiac Magnetic Resonance in Acquired Nonischemic Cardiomyopathies. J Thorac Imaging. 2016 Nov;31(6):348-366. doi: 10.1097/RTI.0000000000000226. PMID 27438188